CLINICAL TRIAL: NCT00536679
Title: An Open Label, Randomised, Single Dose, Three-way Crossover Study to Investigate the Relative Bioavailability of Two Different Formulations of GSK163090 and the Effect of Food on the Pharmacokinetics of a Tablet Formulation in Healthy Male and Female Volunteers
Brief Title: Relative Bioavailability and Food Effect Study for GSK163090 in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 103268
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder and Anxiety Disorders
Keywords: Relative Bioavailability; Randomised; GSK163090; Food Effect
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — 1-(3-(2-(4-(2-methyl-5-quinolinyl)-1-piperazinyl)ethyl)phenyl)-2-imidazolidinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence ABC (Experimental): Subjects will be randomized to sequence ABC, where A=1 milligram (mg) GSK163090 Capsule, Fasted, B=1 mg GSK163090 Tablet, Fasted and C=1 mg GSK163090 Tablet, Fed. In each of the 3 treatment periods, subjects will receive a single oral dose of GSK163090 in the fed or fasted state, followed by a 7-day wash-out period between each dose.
  Interventions: Drug: GSK163090 capsule, fasted; Drug: GSK163090 Tablet, fasted; Drug: GSK163090 Tablet, fed
- Sequence ACB (Experimental): Subjects will be randomized to sequence ACB, where A=1 mg GSK163090 Capsule, Fasted, B=1 mg GSK163090 Tablet, Fasted and C=1 mg GSK163090 Tablet, Fed. In each of the 3 treatment periods, subjects will receive a single oral dose of GSK163090 in the fed or fasted state, followed by a 7-day wash-out period between each dose.
  Interventions: Drug: GSK163090 capsule, fasted; Drug: GSK163090 Tablet, fasted; Drug: GSK163090 Tablet, fed
- Sequence BAC (Experimental): Subjects will be randomized to sequence BAC, where A=1 mg GSK163090 Capsule, Fasted, B=1 mg GSK163090 Tablet, Fasted and C=1 mg GSK163090 Tablet, Fed. In each of the 3 treatment periods, subjects will receive a single oral dose of GSK163090 in the fed or fasted state, followed by a 7-day wash-out period between each dose.
  Interventions: Drug: GSK163090 capsule, fasted; Drug: GSK163090 Tablet, fasted; Drug: GSK163090 Tablet, fed
- Sequence BCA (Experimental): Subjects will be randomized to sequence BCA, where A=1 mg GSK163090 Capsule, Fasted, B=1 mg GSK163090 Tablet, Fasted and C=1 mg GSK163090 Tablet, Fed. In each of the 3 treatment periods, subjects will receive a single oral dose of GSK163090 in the fed or fasted state, followed by a 7-day wash-out period between each dose.
  Interventions: Drug: GSK163090 capsule, fasted; Drug: GSK163090 Tablet, fasted; Drug: GSK163090 Tablet, fed
- Sequence CAB (Experimental): Subjects will be randomized to sequence CAB, where A=1 mg GSK163090 Capsule, Fasted, B=1 mg GSK163090 Tablet, Fasted and C=1 mg GSK163090 Tablet, Fed. In each of the 3 treatment periods, subjects will receive a single oral dose of GSK163090 in the fed or fasted state, followed by a 7-day wash-out period between each dose.
  Interventions: Drug: GSK163090 capsule, fasted; Drug: GSK163090 Tablet, fasted; Drug: GSK163090 Tablet, fed
- Sequence CBA (Experimental): Subjects will be randomized to sequence CBA, where A=1 mg GSK163090 Capsule, Fasted, B=1 mg GSK163090 Tablet, Fasted and C=1 mg GSK163090 Tablet, Fed. In each of the 3 treatment periods, subjects will receive a single oral dose of GSK163090 in the fed or fasted state, followed by a 7-day wash-out period between each dose.
  Interventions: Drug: GSK163090 capsule, fasted; Drug: GSK163090 Tablet, fasted; Drug: GSK163090 Tablet, fed

INTERVENTIONS:
Drug: GSK163090 capsule, fasted — GSK163090 will be available as 1 mg hard gelatine white/white opaque capsules. Each subject will receive a single, oral dose of the study medication on the morning of Day 1. The study drug will be administered with approximately 240 milliliters (mL) of water.
  Other Names: GSK163090
Drug: GSK163090 Tablet, fasted — GSK163090 will be available as 1 mg white coated round tablet. Each subject will receive a single, oral dose of the study medication on the morning of Day 1. The study drug will be administered with approximately 240 mL of water.
Drug: GSK163090 Tablet, fed — GSK163090 will be available as 1 mg white coated round tablet. Each subject will receive a single, oral dose of the study medication on the morning of Day 1. The study drug will be administered with Food and Drug Administration (FDA) high fat breakfast.

SUMMARY:
The study will consist of a screening period, 3 treatment periods and a post-treatment follow-up. In each of the 3 treatment periods, subjects will receive a single oral dose of GSK163090 in the fed or fasted state, followed by a 7-day wash-out period between each dose

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between the ages of 18 and 55 years inclusive.
* If female, the subject is eligible to enter and participate in this study if she is not lactating and is of Non-childbearing potential or
* Child-bearing potential, has a negative pregnancy test at both screen and baseline and agrees to adequate contraception:
* Body weight ≥ 50 kg and body mass index (BMI) between 18.5 - 29.9 kg/m2 inclusive.
* Capable of giving informed consent and can comply with the study requirements and timetable.
* Self-administered Beck Depression Inventory II scale total score no greater than 9, and suicide question score of zero.
* The subject must be able to read, comprehend and record information.
* A signed and dated written informed consent is obtained from the subject.
* Non-smoker (abstinence from smoking for at least 6 months before the start of the study).
* Agrees to abstain from ingesting caffeine or xanthine-containing products for 24 hours prior to the start of dosing until collection of the final pharmacokinetic sample.
* Agree to abstain from alcohol for 24 hours prior to the start of dosing until collection of the final pharmacokinetic sample

Exclusion Criteria:

* As a result of any of the medical interview, physical examination or screening investigations the physician responsible considers the subject unfit for the study.
* The subject has a history of a drug or other allergy which in the opinion of the physician responsible contraindicates their participation in the study.
* The subject is currently participating or has participated in a clinical trial with a new chemical entity during the previous 4 months or any other trial during the previous 3 months.
* The subject has a screening ECG with values outside of protocoled ranges
* The subject has a pulse rate <45 or >100 bpm and a systolic blood pressure >150 and <90 and a diastolic blood pressure >90 and <50.
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* The subject has liver function tests (LFT) elevated >1.5 times above the reference range at pre-study screening that remain elevated with a repeat LFT.
* Any other clinically significant laboratory abnormality.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Abuse of alcohol defined as an average weekly intake of greater than 21 units for males and 14 units for females or an average daily intake of greater than 3 units for males and 2 units for females. 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* Consumption of grapefruit juice or grapefruit within 7 days prior to the first dose of study medication until collection of the last PK sample.
* The subject is unable to abstain from strenuous physical activity for 48 h prior to screening and follow up and for 48 h prior to and 48 h after each treatment period.
* Where participation in study would result in donation of blood in excess of 500 mL within a 90 day period
* An unwillingness of male subjects to abstain from, or use adequate contraception during, sexual intercourse with pregnant or lactating women from the time of the first dose of study medication until 90 days following administration of the last dose of study medication OR An unwillingness of the male subject to use a adequate contraception in addition to having their female partner use another form of contraception if the woman could become pregnant from the time of the first dose of study medication until 90 days following administration of the last dose of study medication.
* Current or recent (within one year) gastrointestinal disease; a history of malabsorption, esophageal reflux, irritable bowel syndrome; frequent (more than once a week) occurrence of heartburn; or any surgical intervention (e.g., cholecystectomy) which would be expected to influence the absorption of drugs.
* The subject has a history of psychiatric illness
* Any history of suicidal attempts or behavior.
* The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen.
* The subject has tested positive for HIV.
* The subject has a past history of drug abuse or has tested positive for urine drugs of abuse at pre-study screening.
* The subject has any history of serotonin syndrome.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09-20 (Actual); Primary Completion 2007-11-05 (Actual); Study Completion 2007-11-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters for GSK163090. Pharmacokinetic blood samples will be collected up to 72 hours post-dose following each dosing session. | 72 hours post-dose following each dosing session.

SECONDARY OUTCOMES:
Additional pharmacokinetic parameters, safety, and tolerability. | 72 hours post-dose following each dosing session.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Neuss, North Rhine-Westphalia, Germany

REFERENCES:
- See also: Results for study 103268 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/103268?search=study&search_terms=103268#rs